CLINICAL TRIAL: NCT02225665
Title: A Phase 1/2, Open-Label Study to Assess the Safety and Tolerability of Repeat Doses of Autologous T-Cells Genetically Modified at the CCR5 Gene by Zinc Finger Nucleases in HIV-Infected Subjects Following Cyclophosphamide Conditioning
Brief Title: Repeat Doses of SB-728mR-T After Cyclophosphamide Conditioning in HIV-Infected Subjects on HAART
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sangamo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SB-728mR-1401
Record Dates: First submitted 2014-08-22; First posted 2014-08-26 (Estimated); Results first posted 2021-02-09 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2020-12

CONDITIONS: Human Immunodeficiency Virus (HIV)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental)
  Interventions: Genetic: SB-728mR-T; Drug: Cyclophosphamide
- Cohort 2 (Experimental)
  Interventions: Genetic: SB-728mR-T; Drug: Cyclophosphamide

INTERVENTIONS:
Genetic: SB-728mR-T — -SB-728mR-T infusions of 2 equal doses 14 days apart (total of up to 40 billion ZFN modified T-cells)
  Arms: Cohort 1
Genetic: SB-728mR-T — - SB-728mR-T infusions of 3 equal doses 14 days apart (total of up to 40 billion ZFN modified T-cells)
  Arms: Cohort 2
Drug: Cyclophosphamide — - IV cyclophosphamide 1 g/m2 two days prior to the first SB-728mR-T infusion

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of repeat doses of T-cell immunotherapy (SB-728mR-T) following cyclophosphamide conditioning.

CCR5 is a major co-receptor for HIV entry into T-cells. Disruption of CCR5 by zinc finger nuclease (SB-728mR), blocks HIV entry into the T-cells, therefore, protects the T-cells from HIV infection. Safety (primary outcome) and anti-viral effect (secondary outcome) of zinc finger nuclease-mediated CCR5 disrupted autologous T-cells (SB-728mR-T) will be evaluated in the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older with documented HIV diagnosis.
* Must be willing to comply with study-mandated evaluations; including discontinuation of current antiretroviral therapy during the treatment interruption.
* Initiated HAART therapy within (≤) 1 year of HIV diagnosis or suspected infection.
* Undetectable HIV-1 RNA for at least 2 months prior to screening and at screening.
* CD4+ T-cell count ≥500 cells/µL.
* Absolute neutrophil count (ANC) ≥ 2500/mm3.
* Platelet count ≥ 200,000/mm3.

Exclusion Criteria:

* Acute or chronic hepatitis B or hepatitis C infection.
* Active or recent (in prior 6 months) AIDS defining complication.
* Any cancer or malignancy within the past 5 years, with the exception of successfully treated basal cell or squamous cell carcinoma of the skin or low grade (0 or 1) anal or cervical dysplasia.
* Current diagnosis of NYHA grade 3 or 4 CHF, uncontrolled angina or uncontrolled arrhythmias.
* History or any features on physical examination indicative of a bleeding diathesis.
* Received HIV experimental vaccine within 6 months prior to screening, or any previous gene therapy using an integrating vector.
* Use of chronic corticosteroids, hydroxyurea, or immunomodulating agents within 30 days prior to screening.
* Use of Aspirin, dipyridamole, warfarin or any other medication that is likely to affect platelet function or other aspects of blood coagulation during the 2 week period prior to leukapheresis.
* Currently participating in another clinical trial or participation in such a trial within 30 days prior to screening visit.
* Currently taking maraviroc or have received maraviroc within 6 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - San Francisco, California
  - Norwalk, Connecticut
  - Orlando, Florida
  - Austin, Texas
  - Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: SB-728mR-T infusions of 2 equal doses 14 days apart (total of up to 40 billion ZFN modified T-cells)
  Cyclophosphamide: - IV cyclophosphamide 1 g/m2 two days prior to the first SB-728mR-T infusion
- Cohort 2: SB-728mR-T infusions of 3 equal doses 14 days apart (total of up to 40 billion ZFN modified T-cells)
  Cyclophosphamide: - IV cyclophosphamide 1 g/m2 two days prior to the first SB-728mR-T infusion
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 3 | 5
Completed | 2 | 4
Not Completed | 1 | 1
Not completed — Subject moved from area and finds it difficult to return for visits. | 1 | 0
Not completed — Subject restarted HAART prior to month 18. | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (8.19) | 39.6 (10.09) | 46.9 (13.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome Measure
Description: Number of Participants with Treatment related Adverse Events in subjects who received any portion of the SB-728mR-T infusion
Time Frame: 12 months
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 5
Participants | 1 | 2

2. Secondary Outcome: Secondary Outcome Measure
Description: Effect of repeat doses of SB-728mR-T on engraftment following cyclophosphamide conditioning as measured by CCR5 Modified CD4 Cells at Month 12.
Time Frame: 12 months
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells 10^9/L
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 2 | 5
cells 10^9/L | 0.090 (0.0015) | 0.162 (0.0818)

3. Secondary Outcome: Secondary Outcome Measure
Description: Effect of SB-728mR-T on plasma HIV-1 RNA levels following HAART interruption
Time Frame: 12 months
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: log copies/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 2 | 5
log copies/mL | 3.218 (1.9243) | 1.228 (1.7029)

4. Secondary Outcome: Secondary Outcome Measure
Description: Change from baseline to month 12 in CD4+ T-cell counts in peripheral blood after repeat treatments with SB-728mR-T. (i.e. month 12 value - baseline value)
Time Frame: Baseline and 12 months
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells 10^9/L
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 2 | 5
cells 10^9/L | -0.178 (0.0445) | 0.078 (0.2796)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=5)
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Chlamydial infection (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 | 2
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All proposed written materials related to the study or an outline of any proposed oral presentations, shall be submitted to Sangamo for approval at least 45 days prior to submission of materials for publication or any oral disclosure to a third party. If Sangamo determines that a description of patentable subject matter is contained in such written material or outline, it shall notify the clinical site within 1 month after receipt and Sangamo will have an additional 90 days for review.

DOCUMENTS (3):
  • Study Protocol: Protocol Amendment 2 Signature page (2014-10-15): https://cdn.clinicaltrials.gov/large-docs/65/NCT02225665/Prot_000.pdf
  • Study Protocol: Protocol Amendment 2 (2014-10-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT02225665/Prot_001.pdf
  • Statistical Analysis Plan (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/65/NCT02225665/SAP_002.pdf